CLINICAL TRIAL: NCT04634162
Title: Pharmacodynamic and Pharmacokinetic Profiles of Switching Between Cangrelor and Ticagrelor Following Ticagrelor Pre-treatment: The Switching Antiplatelet -5 (SWAP-5) Study
Brief Title: PD and PK Profiles of Switching Between Cangrelor and Ticagrelor Following Ticagrelor Pre-treatment
Acronym: SWAP-5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Scott R. MacKenzie Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMF-01
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: ticagrelor; cangrelor; switching
MeSH Terms: conditions — Coronary Artery Disease | interventions — cangrelor; Saline Solution

STUDY DESIGN:
Intervention Model Description: The Switching Antiplatelet Therapy-5 (SWAP-5) study will be a prospective, randomized, double-blind, placebo controlled, cross-over PK and PD investigation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, research staff and laboratory personnel will be blinded to treatment assignments. Masking and randomization of medications (cangrelor and placebo) will be performed by our institutional research pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cangrelor (Experimental): Ticagrelor loading dose followed after 1 hour by cangrelor bolus and infusion
  Interventions: Drug: Cangrelor; Drug: Placebo
- Placebo (Placebo Comparator): Ticagrelor loading dose followed after 1 hour by placebo infusion
  Interventions: Drug: Cangrelor; Drug: Placebo

INTERVENTIONS:
Drug: Cangrelor — Cangrelor will be used at the FDA recommended dose using a 30 μg/kg bolus followed by 4 μg/kg/min infusion. The duration of cangrelor/placebo infusion will be 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase
  Other Names: Kengreal
Drug: Placebo — Normal saline will be infused for 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase
  Other Names: Normal saline

SUMMARY:
Cangrelor is an intravenous P2Y12 inhibitor utilized as a bridge to achieve adequate platelet inhibition until oral P2Y12 inhibitors achieve their full antiplatelet effects in patients undergoing coronary stenting. Although in this setting the potent oral P2Y12 inhibitor ticagrelor is commonly utilized, there is very limited data on the optimal approach for switching between these therapies. The methodological approach for this assessment should rely on comprehensive pharmacodynamics (PD) investigations aimed to assess levels of P2Y12 receptor inhibition, pharmacokinetic (PK) investigations to assess systemic levels of the drug/drug metabolite, and mechanistic investigations by assessment of levels of P2Y12 receptor gene expression. The overarching aim of this investigation is to rule out a drug-drug interaction when ticagrelor is administered prior to cangrelor infusion.

DETAILED DESCRIPTION:
Cangrelor is an intravenous P2Y12 inhibitor utilized as a bridge to achieve adequate platelet inhibition until oral P2Y12 inhibitors achieve their full antiplatelet effects in patients undergoing coronary stenting. Although in this setting the potent oral P2Y12 inhibitor ticagrelor is commonly utilized, there is very limited data on the optimal approach for switching between these therapies. In particular, ruling out a drug-drug interaction (DDI) is critical to this extent as the presence of a DDI would translate into reduced or abolished antiplatelet effects exposing these acute patients to an increased thrombotic risk. Despite the available evidence suggesting a lack of DDI with the use of ticagrelor in cangrelor treated patients, most data derive from studies in which ticagrelor was given at the time of initiation or during cangrelor infusion. To date, there is no data to fully rule out a DDI when ticagrelor is given prior to starting cangrelor infusion. The need for such investigation is underscored by the relatively high prevalence of pretreatment with ticagrelor in acute settings. The methodological approach for this assessment should rely on comprehensive pharmacodynamics (PD) investigations aimed to assess levels of P2Y12 receptor inhibition, pharmacokinetic (PK) investigations to assess systemic levels of the drug/drug metabolite, and mechanistic investigations by assessment of levels of P2Y12 receptor gene expression. The overarching aim of this investigation is to rule out a DDI when ticagrelor is administered prior to cangrelor infusion.

ELIGIBILITY:
Inclusion criteria:

* Patients with known coronary artery disease (defined as prior type I myocardial infarction, coronary revascularization, percutaneous or surgical, or presence of at least a 50% stenosis in any major epicardial vessel).
* Age > 18 years old
* On aspirin 81mg/qd for at least 1 month

Exclusion criteria:

* Inability to provide written informed consent
* Hemodynamic instability
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in past 30 days
* Known allergies to ticagrelor or cangrelor
* Considered at high risk for bleeding
* History of intracranial bleeding/hemorrhagic stroke
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban, apixaban, edoxoban) within past 30 days
* Known platelet count <80x106/mL
* Known hemoglobin <10 g/dL
* Active bleeding
* Known end stage renal disease on hemodialysis
* Known severe hepatic dysfunction
* Acute or severe bronchial asthma or upper airway obstruction.
* Patients with sick sinus syndrome (SSS) or high degree AV block without pacemaker protection.
* Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with ticagrelor): Ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromizycin.
* Pregnant females [women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Franchi, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share study data

REFERENCES:
- [Derived] Franchi F, Ortega-Paz L, Rollini F, Galli M, Been L, Ghanem G, Shalhoub A, Ossi T, Rivas A, Zhou X, Pineda AM, Suryadevara S, Soffer D, Zenni MM, Reiter B, Jilma B, Angiolillo DJ. Cangrelor in Patients With Coronary Artery Disease Pretreated With Ticagrelor: The Switching Antiplatelet (SWAP)-5 Study. JACC Cardiovasc Interv. 2023 Jan 9;16(1):36-46. doi: 10.1016/j.jcin.2022.10.034. Epub 2022 Oct 31. PMID 36317958

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 22 patients were consented and enrolled in the study: 2 patients were eligible for randomization due to the presence of exclusion criteria. A total of 20 patients were randomized and exposed to at least one dose of study medication.
Groups:
- Cangrelor First, Then Placebo: icagrelor loading dose followed after 1 hour by cangrelor bolus and infusion Cangrelor: Cangrelor will be used at the FDA recommended dose using a 30 μg/kg bolus followed by 4 μg/kg/min infusion. The duration of cangrelor/placebo infusion will be 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase.
  Placebo: Normal saline will be infused for 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase.
- Placebo First, Then Cangrelor: Ticagrelor loading dose followed after 1 hour by placebo infusion Cangrelor: Cangrelor will be used at the FDA recommended dose using a 30 μg/kg bolus followed by 4 μg/kg/min infusion. The duration of cangrelor/placebo infusion will be 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase.
  Placebo: Normal saline will be infused for 2 hours. After completing the first phase of the study, patients will undergo a 1-4 week wash-out period and then will cross-over to the alternative treatment in the second phase.
Period: Phase 1 Pre-cossover
Arm/Group | Cangrelor First, Then Placebo | Placebo First, Then Cangrelor
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Phase 2 Post-cossover
Arm/Group | Cangrelor First, Then Placebo | Placebo First, Then Cangrelor
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Whole Study Population: Using a computer-based randomization system, patients were randomly assigned in a 1:1 fashion to 1 of the following treatment arms: 1) ticagrelor loading dose (LD) followed after 1 hour by cangrelor bolus and infusion; or 2) ticagrelor LD followed after 1 hour by placebo bolus and infusion. Ticagrelor was administered as a 180-mg LD and cangrelor as a 30-μg/kg bolus followed by 4-μg/kg/min infusion. Cangrelor/placebo infusion was continued for a duration of 2 hours. After completing the first phase of the study, patients underwent a 1- to 4-week washout period and then crossed over to the alternative treatment in the second phase (ie, patients assigned to treatment with cangrelor in the first phase were assigned to placebo in the second phase and vice versa).
Arm/Group | Whole Study Population
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20
Prior myocardial infatction [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Platelet Reactivity Measured by VerifyNow
Description: The primary end point of the study will be the non-inferiority in P2Y12 reaction units (PRU) measured by VerifyNow after discontinuation of cangrelor vs. placebo
Time Frame: 2 hours
Measure: Least Squares Mean (Inter-Quartile Range); unit: P2Y12 reaction units
Arm/Group | Cangrelor | Placebo
Number analyzed (Participants) | 20 | 20
P2Y12 reaction units | 16.9 [-11.8 to 45.7] | 12.6 [-16.1 to 41.4]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Cangrelor | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 9/20 | 9/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cangrelor (N=20) | Placebo (N=20)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 9 (9) — Shortness of breath

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04634162/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/62/NCT04634162/ICF_001.pdf